CLINICAL TRIAL: NCT03220503
Title: Effect of Endometrial Injury Before Frozen Embryo Transfer on Pregnancy Rate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Yasser sherbiny, Principal Investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AinShamsMH Ysherbiny
Record Dates: First submitted 2017-06-15; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) (Experimental): consists of 25 patients will receive frozen embryo with endometrial scratching on day 7 of transfer cycle.
  Interventions: Procedure: endometrial injury
- Group (B) (No Intervention): consists of 25 patients will receive frozen embryo without endometrial scratching as control group.

INTERVENTIONS:
Procedure: endometrial injury — single induced injury will be done on the posterior endometrium on day 7 of the transfer cycle by using modified Cook catheter.
  Arms: Group (A)

SUMMARY:
Research Question:

In women undergoing frozen embryo transfer, does routine endometrial injury before frozen embryo transfer increase clinical pregnancy rate?

Research Hypothesis:

(Null Hypothesis) In women undergoing frozen embryo transfer Routine endometrial injury before frozen embryo transfer does not increase clinical pregnancy rate.

(Alternative Hypothesis) In women undergoing frozen embryo transfer, endometrial injury before the transfer may increase pregnancy rate.

DETAILED DESCRIPTION:
Suitable women will be invited to participate in the study then a signed and informed consent will be obtained from them. When the patient's consent is obtained, they are to be included into the study.

Data Collection:

During first visit, all patients will undergo complete clinical examination and detailed medical history will be obtained. Each patient will have a Case Record Form (CRF) in which the following data will be recorded.

* Patient number (according to the randomization schedule).
* Age, BMI.
* Past medical and surgical history.
* Duration of infertility.

Procedure:

Endometrial injury:

A single induced injury will be done on the posterior endometrium on day 7 of the transfer cycle by using modified Cook catheter Protocol for vitrification Embryos will first loaded with equilibrium solution containing7.5% ethylene glycol (EG) and 7.5% dimethyl sulphoxide (DSMO) (Sigma-Aldrich) for 5-10 minute at room temperature and then with vitrification solution containing 15% EG, 15% DSMO and 0.5 mol/L sucrose for 50-60 seconds at room temperature. After observed cellular shrinkage, embryos will quickly stored in liquid nitrogen (LN) for at least 2 months. At warming, embryos will removed from LN and embryos will exposed to thawing solution containing sucrose at 37°C temperature for 50-60 seconds and then embryos will sequentially incubated in diluents solutions before being transferred .

Evaluation and transfer of thawed embryos After thawing, each embryo will evaluated twice, once immediately for the number of surviving blastomeres and again after 18 hours post-thaw in vitro culture for assessing of mitosis and number of blastomeres. Embryos will considered survived if >50% of each blastomere are intact and selected for intrauterine transfer (Depending on patients' embryos, 2 or 3 embryos will transferred).

Embryos will classified as fully intact or excellent morphology (100% cells survived with <10% fragmentation) or good morphology (100% cells survived with 10%-20% fragmentation), partially damaged or poor morphology (≥50% cells survived with or without any fragmentation) and Degenerated embryos (<50% cells survived) .Only fully intact and partially damaged embryos will transferred. Degenerated or arrested embryos will not transferred.

Protocol of endometrial preparation before Frozen Embryo Transfer (FET) :

There are different protocols for FET cycles. That is true for both "natural cycle" FETs and for "hormone replacement cycle" frozen-thawed embryo transfers. We will use hormone replacement cycles because they have better success rates. However, some clinics offer a natural cycle FET approach. Success rates are higher with hormone replacement, or "controlled" FET cycles.

Medicines and Drugs in a Frozen Embryo Transfer FET Cycle

1. Gonadotropin-Releasing Hormone agonist (such as Lupron) will be given, either midluteal (day 21) or overlapping with a birth control pill.
2. Down-regulation will be confirmed by ultrasound and blood tests.
3. Estradiol valerate 2 mg twice daily (orally) will start after the period. This dose may need to be increased after monitoring of the uterine lining thickness.
4. When the endometrium has a "good" thickness( > 8 mm), progesterone will be started (intramuscular shots, or a vaginal product).
5. Embryo transfer will be planned for 3-6 days later - depending on the stage of development of the embryos to be transferred.
6. Estrogen and progesterone will be continued in the luteal phase.
7. Pregnancy testing will be done 9-14 days after transfer - depending on the stage of development of the embryos replaced and the preferences of the fertility clinic.
8. If pregnant, estrogen and progesterone will be continued until about 10-15 weeks of pregnancy and then weaned off.

ELIGIBILITY:
Inclusion Criteria:

* All infertile women have high quality frozen embryos.

Exclusion Criteria:

* History of endocrine disease such as: diabetes; Hyperthyroidism and Hyperprolactinemia.
* History of hysteroscopic surgery due to intrauterine adhesions.
* History of cardiovascular, renal or liver disease .
* History of stroke or myocardial infarction.
* Poor quality embryos.
* Alcohol or Substance abuse.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-09-09 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Chemical pregnancy rate | two weeks after frozen embryo transfer
  serum Beta -Human Chorionic Gonadotropin positive

SECONDARY OUTCOMES:
Clinical pregnancy rate | four weeks after frozen embryo transfer
  appearance of gestational sac on trans-vaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Adel Sh Salah El-Din, Ass. Prof., Study Director — Ain Shams University; Mohammed A Faris, Lecturer, Study Director — Ain Shams University; Mohamed E Shawky, Lecturer, Study Director — Ain Shams University
Locations (1):
- ART unit - Ain Shams university Matrnity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided